CLINICAL TRIAL: NCT05866913
Title: Effect of Neurodynamics vs Passive Stretching in Federated Soccer Players With Short Hamstring Syndrome
Brief Title: Neurodynamics vs. Stretching in Soccer Players With Short Hamstring Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Angel Martínez Carrasco, Professor Phd, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FJMG-2023-1
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Hamstring Contractures
Keywords: Peripheral nervous system; Muscle stretching exercises; Hamstring muscles; Sciatic nerve; Elasticity

STUDY DESIGN:
Intervention Model Description: Control group. Experimental group 1. Experimental group 2.
Who Masked: Participant
Masking Description: Only the participants will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): Passive shoulder mobilizations for 90 seconds.
  Interventions: Procedure: passive shoulder mobilization.
- Experimental group 1 (Experimental): Sciatic nerve glide in a seated slump position for 90 seconds.
  Interventions: Procedure: Sciatic nerve slippage.
- Experimental group 2 (Experimental): Passive stretching of the hamstring muscles with straight leg raising for 90 seconds.
  Interventions: Procedure: Passive stretching of the hamstring muscles.

INTERVENTIONS:
Procedure: Sciatic nerve slippage. — Sciatic nerve slippage.
  Arms: Experimental group 1
Procedure: Passive stretching of the hamstring muscles. — Passive stretching of the hamstring muscles.
  Arms: Experimental group 2
Procedure: passive shoulder mobilization. — passive shoulder mobilization.
  Arms: Control group

SUMMARY:
Comparison of the effects of passive stretching vs. sciatic nerve gliding in soccer players presenting with short hamstring syndrome.

DETAILED DESCRIPTION:
Soccer players from three teams in the region of Murcia (Spain) were recruited and randomly divided into three groups: control group, experimental group 1 and experimental group 2.

In the control group passive shoulder mobilization will be applied, in experimental group 1 sciatic nerve gliding will be applied and in experimental group 2 passive hamstring stretching will be applied.

Treatments will be performed once a week for 4 weeks and measurements will be taken at week 1 and 4.

ELIGIBILITY:
Inclusion Criteria:

* Soccer players of the Murcia Region Federation who have short hamstring syndrome.
* Between 16 and 30 years of age.
* To complete the informed consent form.

Exclusion Criteria:

* Subjects with significant neurological pathology.
* Subjects with hamstring muscle injury.
* Subjects with lumbar pathology.

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Elasticity of the hamstring muscles. | One month
  Measurement in degrees of the articular range of the hamstring muscles, using a goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Ángel Martínez Carrasco, PhD, Principal Investigator — Universidad de Murcia
Locations (1):
- Universidad de Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No